CLINICAL TRIAL: NCT05123742
Title: Pragmatic Return to Effective Dental Infection Control Through Triage and Testing (PREDICT): A PBRN Feasibility Study on COVID-19 Screening in Dental
Brief Title: PREDICT: A PBRN Feasibility Study on COVID-19 Screening in Dental Practice
Acronym: PREDICT
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); The National Dental Practice-Based Research Network (Network); Kaiser Foundation Research Institute (Other); University of Alabama at Birmingham (Other); University of Rochester (Other); University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Cecile A. Feldman, DMD, Professor and Dean, Rutgers School of Dental Medicine, Rutgers, The State University of New Jersey
Other Study IDs: Pro2021000968; IRB-300007026 (Other: University of Alabama at Birmingham); U01DE028727 (NIH)
Record Dates: First submitted 2021-10-20; First posted 2021-11-17 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: COVID-19 Infection
Keywords: dental health care; antibody test; antigen test; dental practice environment; COVID-19 screening; point of care testing; lab-based testing; dental offices; pragmatic design
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biospecimens - saliva sample, tongue swab, nasal swab specimen, and capillary blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DHCW Subjects: Dental Health Care Workers
  Interventions: Diagnostic Test: COVID-19 Testing
- Patient Subjects: Dental patients
  Interventions: Diagnostic Test: COVID-19 Testing

INTERVENTIONS:
Diagnostic Test: COVID-19 Testing — Testing for the SARS-CoV-2 virus

SUMMARY:
The study team will conduct a feasibility study to develop and test out procedures for improved triage and COVID-19 testing in dental practices to increase safety and perceptions of the safety of Dental Health Care Workers (DHCW) and their patients. DHCWs in offices with Practice-Based Regional Network (PBRN) members and their patients will be recruited to participate in one of two protocols. The first, point-of-care (POC), will test out procedures for point-of-care SARS-CoV-2 antigen testing in the dental office along with enhanced triage using pulse oximeters. The second, laboratory (LAB), will test out procedures for a saliva-based laboratory SARS-CoV-2 viral test along with enhanced triage. The feasibility of implementing COVID-related testing and enhanced triage procedures in the dental setting will provide preliminary data to inform a larger network-wide study grant application.

DETAILED DESCRIPTION:
Data derived from this research would enable dental health care workers to return to work, providing essential oral health care services in the safest possible environment. It will provide patients with confidence that they could resume seeking dental care under optimal conditions that ensure their well-being. The specific aims of this proposal are divided into three parts. The first aim is to apply the Delphi methodology, selecting a facilitator, a panel of experts, defining the problem, addressing the problem with several iterations, and coming to a consensus solution. The second aim is will address the concerns and recommended solutions proposed by the Delphi group and formulated into pragmatic improvements that can be applied to improved practice procedures that can be formulated into testable hypotheses that can be incorporated into a practice strategy for the future of dentistry. Pragmatic and novel methodological changes developed by the investigative team will be presented once again to the Delphi group to gain their approval and/or recommended modifications. Our overarching goal is to test these "improved" strategies in a pilot study and as such the investigators are looking to incorporate two to three methodological suggestions that can be fit into a pragmatic re-design of "best dental practices". Thus, the third aim is designed to test these "best dental practice" approaches in a pilot study. The goal of the third aim is to evaluate how each of these strategies can be applied to different office settings. The data derived from this approach will be used to provide a sample size calculation for a larger study using the PBRN framework for office participation. The all-encompassing aim of the study is to develop a new way of approaching dental practice that ensures a sense of security and practicality for both patients and health professionals. The hypothesis to be tested derived from these aims relates to the structured development of several methodologies that can be applied to dental practice. These methodologic improvements in dental practice will be based on the most current scientific knowledge that can be applied to ensure safety in a dental office setting. To re-iterate the purpose of this study developed from the three aims proposed is to assess and compare each of the pragmatic models developed such that a sample size calculation can be computed. The pilot study design and the sample size calculation derived from this pilot data will compare two to three pragmatic/innovative modifications in the current practice guidelines and provide an estimate that can utilize the larger PBRN framework to best determine the generalizability of the models chosen for study.

ELIGIBILITY:
Inclusion Criteria:

A Dental Health Care Worker must meet all of the following criteria to be eligible to participate in the study:

* Be 18 years or older
* Be a National Dental PBRN member dentist or work in a dental office with a National Dental PBRN member dentist who consents to study participation
* Be able to understand the informed consent.
* Provide signed and dated informed consent form
* Be able to understand all instructions for data collection instruments
* Be willing and able to comply with all study procedures, including COVID-19 testing, and be available for the duration of the study

A Patient must meet all of the following criteria to be eligible to participate in the study:

* Be 18 years or older
* Be able to understand the informed consent.
* Have a computer or electronic tablet with internet access
* Able to complete consent and questionnaire on a computer or electronic tablet
* Provide signed and dated informed consent form
* Be able to understand all instructions for data collection instruments
* Be willing and able to comply with all study procedures, including having a COVID-19 test performed

Exclusion Criteria:

* Children less than 18 years will not be able to participate.
* Participants would be excluded if they participated in the feasibility study previously conducted at Rutgers University.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female dental health care workers and patients who are seen in a Practice-Based Research Network dentist office.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecile Feldman, DMD, Principal Investigator — Rutgers School of Dental Medicine; Janine Fredericks-Younger, DMD, Principal Investigator — Rutgers School of Dental Medicine; Modupe Coker, PhD, Principal Investigator — Rutgers School of Dental Medicine; Daniel Fine, DMD, Principal Investigator — Rutgers School of Dental Medicine; Gayathri Subramanian, DMD, Principal Investigator — Rutgers School of Dental Medicine; Maria Gennaro, PhD, Principal Investigator — Rutgers University; Cyril Meyerowitz, DDS, Study Director — University of Rochester; Veerasathpurush Allareddy, PhD, Study Director — University of Illinois at Chicago
Locations (1):
- Rutgers School of Dental Medicine, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
If the COVID test results show that a participant is positive for COVID-19, the study staff will tell the participant the results. The study staff will be required to give the participant's name to the state's Department of Public Health if the participant tests positive because this is the law.
  At the end of the study, de-identified data will be provided to the National Coordinating Center.

REFERENCES:
- [Derived] Fredericks-Younger J, Feldman CA, Allareddy V, Funkhouser E, McBurnie M, Meyerowitz C, Ragusa P, Chapman-Greene J, Coker M, Fine D, Gennaro ML, Subramanian G. Pragmatic Return to Effective Dental Infection Control through Triage and Testing (PREDICT): an observational, feasibility study to improve dental office safety. Pilot Feasibility Stud. 2024 Feb 28;10(1):44. doi: 10.1186/s40814-024-01471-x. PMID 38419131
- [Derived] Fredericks-Younger J, Feldman C, Allareddy V, Funkhouser E, McBurnie M, Meyerowitz C, Ragusa P, Chapman-Greene J, Coker M, Fine DH, Gennaro ML, Subramanian G. Pragmatic Return to Effective Dental Infection Control through Triage and Testing (PREDICT): A feasibility study to improve dental office safety. Res Sq [Preprint]. 2023 Sep 7:rs.3.rs-3011647. doi: 10.21203/rs.3.rs-3011647/v1. PMID 37720040
- [Derived] Fredericks-Younger J, Fine DH, Subramanian G, Coker MO, Meyerowitz C, Ragusa P, Allareddy V, McBurnie MA, Funkhouser E, Gennaro ML, Feldman CA. The Pragmatic Return to Effective Dental Infection Control Through Triage and Testing (PREDICT) Study: Protocol for a Prospective Clinical Study in the National Dental Practice-Based Research Network. JMIR Res Protoc. 2022 Aug 31;11(8):e38386. doi: 10.2196/38386. PMID 35944181

RESULTS

PARTICIPANT FLOW:
Groups:
- DHCW - POC: Dental Health Care Workers undergoing point of care testing
- DHCW - LAB: Dental Healthcare Workers undergoing laboratory testing
- Patients - POC: Patients undergoing point of care testing
- Patients - LAB: Patients undergoing laboratory based testing
Period: Overall Study
Arm/Group | DHCW - POC | DHCW - LAB | Patients - POC | Patients - LAB
Started | 13 | 16 | 20 | 23
Completed | 13 | 15 | 19 | 22
Not Completed | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Dental Healthcare Workers - POC: Dental Health Care Workers recruited who work in a participating dental office undergoing point-of-care testing
- Dental Healthcare Workers - LAB: Dental Health Care Workers recruited who work in a participating dental office undergoing lab based testing
- Patient - POC: Patients recruited who work in a participating dental office undergoing point-of-care testing
- Patients-LAB: Patients recruited who work in a participating dental office undergoing lab based testing
- Total: Total of all reporting groups
Arm/Group | Dental Healthcare Workers - POC | Dental Healthcare Workers - LAB | Patient - POC | Patients-LAB | Total
Number analyzed (Participants) | 13 | 16 | 20 | 23 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 17 | 15 | 57
  >=65 years | 1 | 3 | 3 | 8 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 14 | 13 | 51
  Male | 2 | 3 | 6 | 10 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 6 | 0 | 9
  Not Hispanic or Latino | 8 | 15 | 14 | 22 | 59
  Unknown or Not Reported | 3 | 0 | 0 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 2
  White | 10 | 15 | 18 | 20 | 63
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 2 | 1 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Perception of Safety
Description: Participants perception of safety in the dental office. Outcome measure is a score on a scale from 0 to 100 where 0=has unsafe as one can possibly feel and 100=as safe as one can possibly feel. All participants (DHCW and patients) were asked to indicate how safe they would feel seeking dental care if all dental office workers, but not patients, were regularly tested: how safe they would feel seeking care if all patients, but not dental care workers, were tested prior to their dental appointments; and how safe they would feel seeking dental care if all dental workers were regularly tested AND all patients were tested prior to their dental appointments.
Time Frame: For DHCW at Day 28 (+/- 14 days), For Patients at their dental visit (day 1)
Population: Only participants who completed the protocol have been included in the analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Patients-POC: Patients participating in study undergoing point of care testing
- Dental Healthcare Workers - POC: Dental Healthcare Workers participating in study undergoing point of care testing
- Dental Healthcare Workers - LAB: Dental Healthcare Workers undergoing LAB testing
- Patients - LAB: Patients participating in study undergoing laboratory based testing
Arm/Group | Patients-POC | Dental Healthcare Workers - POC | Dental Healthcare Workers - LAB | Patients - LAB
Number analyzed (Participants) | 19 | 13 | 15 | 22
score on a scale
  Perception of safety when only patients are tested | 60 [29 to 98] | 74 [50 to 85] | 51 [48 to 76] | 52.5 [37 to 65]
  Perception of safety when only DHCW are tested | 95 [80 to 100] | 82 [73 to 90] | 60 [50 to 83] | 71 [62 to 76]
  Perception of safety when both patients and DHCW are tested | 100 [94 to 100] | 96 [89 to 100] | 75 [52 to 86] | 93 [82 to 100]

2. Secondary Outcome: Specimen Preference
Description: Ranking of the type of specimen participants preferred. Outcome measure is a score on a scale from 1 to 6 where 1=the most preferred specimen type and 6 the least preferred specimen type. Scores could not be used twice providing a ranking of specimen preference.
Time Frame: For DHCWs at Day 28 (+/- 13 days); For patients at the time of their dental visit (Day 1)
Population: Analysis population is limited to those participants who completed the protocol
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- DHCW - :LAB: Dental Healthcare Workers undergoing laboratory based testing
- Patient - LAB: Patients undergoing laboratory based testing
Arm/Group | DHCW - POC | DHCW - :LAB | Patients - POC | Patient - LAB
Number analyzed (Participants) | 13 | 15 | 19 | 22
score on a scale
  Saliva | 1 [1 to 3] | 2 [1 to 2] | 3 [1 to 4] | 2 [1 to 2]
  Tongue Epithelial Cells | 2 [1 to 3] | 2 [1 to 2] | 2 [1 to 3] | 2 [1 to 3]
  Nasal Swab | 2 [1 to 3] | 3 [2 to 3] | 1 [1 to 3] | 2 [2 to 3]
  Nasal-Pharyngeal Swab | 4 [3 to 4] | 4 [4 to 4] | 6 [2 to 6] | 4 [4 to 4]
  Finger Stick (Capillary Blood) | 5 [5 to 5] | 5 [5 to 5] | 5 [3 to 6] | 5 [5 to 5]
  Venous Blood | 6 [6 to 6] | 6 [6 to 6] | 6 [5 to 6] | 6 [6 to 6]

3. Secondary Outcome: Testing Protocol Preference
Description: COVID-19 testing method preferred by subjects. Outcomes measure is a score on a scale where testing protocols are ranking from 1 to 4 with 1 being the most preferred method and 4 is the least preferred method. Score could not be used twice with the scores indicating the subject's testing preference.
Time Frame: For DHCWs at Day 28 (+/- 14 days); For Patients at time of their dental visit (Day 1)
Population: Only participants who completed the protocol are included in this analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- DHCW - LAB: Dental Healthcare Workers undergoing laboratory based testing
Arm/Group | DHCW - POC | DHCW - LAB | Patients - POC | Patients - LAB
Number analyzed (Participants) | 13 | 15 | 19 | 22
score on a scale
  Specimen collected at home and mailed to the lab for processing | 2 [2 to 4] | 1 [1 to 2] | 2 [1 to 2] | 1 [1 to 2]
  Point-of-care test in the dental office | 1 [1 to 2] | 3 [1 to 3] | 2 [1 to 3] | 2.5 [1 to 3]
  Specimen collected in the dnetal office and mail to the lab for processing | 3 [2 to 3] | 2 [2 to 2] | 3 [3 to 3] | 2 [2 to 3]
  Specimen collected at a commercial lab and processed at the lab | 4 [3 to 4] | 4 [4 to 4] | 4 [3 to 4] | 4 [4 to 4]

ADVERSE EVENTS:
Time Frame: For DHCWS - 28 days +/- 14 days: For patients 1 day
Groups:
- DHCW - POC: Dental healthcare workers participating in the point-of-care protocol
- DHCW - LAB: Dental healthcare workers participating in the laboratory based protocol
- Patients - POC: Patients participating in the POC protocol
- Patients - LAB: Patients participating in the LAB protocol
Arm/Group | DHCW - POC | DHCW - LAB | Patients - POC | Patients - LAB
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/15 | 0/19 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15 | 0/19 | 0/22
Other Adverse Events (participants affected / at risk) | 0/13 | 0/15 | 0/19 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT05123742/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT05123742/ICF_000.pdf